CLINICAL TRIAL: NCT03827564
Title: Goblet Cell Degranulation Produced by Nasal Neurostimulation: A Randomized, Controlled Study in Patients With Dry Eye Disease
Brief Title: Goblet Cell Degranulation Produced by Intranasal Tear Neurostimulator (ITN) in Dry Eye Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study discontinued due to business reasons.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1919-802-019
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ITN [TrueTear®] - Intranasal Application (Experimental): Intranasal application of the ITN. Single application at application visit.
  Interventions: Device: Intranasal Tear Neurostimulator (ITN) [TrueTear®]
- ITN [TrueTear®] - Extranasal Application (Experimental): Extranasal application of the ITN. Single application at application visit.
  Interventions: Device: Intranasal Tear Neurostimulator (ITN) [TrueTear®]

INTERVENTIONS:
Device: Intranasal Tear Neurostimulator (ITN) [TrueTear®] — The ITN applies a small electrical current to the nasal cavities to gently activate the body's natural tear production system.

SUMMARY:
The purpose of this study is to evaluate goblet cell degranulation following acute use of the Intranasal Tear Neurostimulator in participants with dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving verbal and signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol
* Have not worn contact lenses for at least 7 days prior to the screening visit and are willing to forego the use of contact lenses for the duration of the study
* The participant should be literate, able to speak English, and able to complete questionnaires independently

Exclusion Criteria:

* Chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the investigator, may lead to clinically significant increased bleeding
* Nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
* Cardiac demand pacemaker, implanted defibrillator or other implanted electronic device
* Corneal transplant in either or both eyes
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
* Women who are pregnant, planning a pregnancy, or nursing throughout the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pflugfelder, MD, Principal Investigator — Baylor College of Medicine, Department of Ophthalmology
Locations (1):
- Baylor College of Medicine - Department of Ophthalmology, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, SAP
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ITN [TrueTear®] - Intranasal Application | ITN [TrueTear®] - Extranasal Application
Started | 9 | 5
Completed | 8 | 5
Not Completed | 1 | 0
Not completed — Discontinued due to Study Termination | 1 | 0

BASELINE CHARACTERISTICS:
Population: All 14 enrolled participants were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | ITN [TrueTear®] - Intranasal Application | ITN [TrueTear®] - Extranasal Application | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (15.4) | 46.8 (10.4) | 52.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Ratio of Degranulated Goblet Cells.
Description: Mean change from Screening to Application Visit in ratio of goblet cell degranulation post-intranasal use of the Intranasal Tear Neurostimulator (ITN) at the Application visit compared to without use of the ITN at the Screening visit
Time Frame: Screening (Day -60 to Day -30) to Application Visit (Day 0)
Population: Of the 14 Randomized participants, 13 received a single application of the Intranasal Tear Neurostimulator (ITN)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | ITN [TrueTear®] - Intranasal Application | ITN [TrueTear®] - Extranasal Application
Number analyzed (Participants) | 6 | 5
Ratio | 0.007 (0.171) | 0.124 (0.069)

ADVERSE EVENTS:
Time Frame: Adverse data was collected from participants at Screening (Day -60 to Day -30) to the Application Visit (Day 0), with a 30-day safety follow-up after the application. A period of 60 to 90 days in total.
Arm/Group | ITN [TrueTear®] - Intranasal Application | ITN [TrueTear®] - Extranasal Application
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/5

LIMITATIONS AND CAVEATS:
This study was terminated early, resulting in a small number of patients analyzed. Only a descriptive statistical analysis will be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Allergan as the sponsor has proprietary interest in this study. Authorship and manuscript composition will reflect joint cooperation between investigators and Allergan personnel. Authorship will be established prior to the writing of the manuscript. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT03827564/Prot_000.pdf